CLINICAL TRIAL: NCT02682485
Title: A Multicenter, Phase II, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial of Serial Endoscopic Surveillance (SES) and Direct Topical Antibiotics (DTA) to Define the Role of Microbes in Anastomotic Healing
Brief Title: Serial Endoscopic Surveillance & Direct Topical Antibiotics to Define the Role of Microbes in Anastomotic Healing
Acronym: SES-DTA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB15-0971
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Anastomotic Leak; Rectal Cancer
Keywords: Rectal Cancer; low anterior resection; SES; SES-DTA; anastomotic leak; anastomotic healing; intestinal healing; anastomosis
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms | interventions — Ciprofloxacin; Metronidazole; Neomycin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cipro, metronidazole, neomycin combo (Experimental): As part of each serial endoscopic surveillance, a second lavage of the anastomosis will be performed prior to removing the endoscope. In this arm, the lavage will be with a direct topical antibiotics solution composed of metronidazole, ciprofloxacin and neomycin.
  Interventions: Drug: Cipro, metronidazole, neomycin combo; Procedure: Serial Endoscopic Surveillance
- Saline (Placebo Comparator): As part of each serial endoscopic surveillance, a second lavage of the anastomosis will be performed prior to removing the endoscope. In this arm, the lavage will be with direct topical saline.
  Interventions: Procedure: Serial Endoscopic Surveillance; Drug: Saline

INTERVENTIONS:
Drug: Cipro, metronidazole, neomycin combo — During endoscopies after imaging, the anastomosis will be lavaged with an antibiotic solution composed of metronidazole, ciprofloxacin and neomycin
  Other Names: Cipro/CiproXR/CiproIV; Flagyl/FlagylER/Metro; Neomycin
  Arms: Cipro, metronidazole, neomycin combo
Procedure: Serial Endoscopic Surveillance — Patients will undergo serial endoscopic surveillance consisting of three endoscopies: one intra-operative endoscopy (POD0) and two post-operative endoscopies (POD3-7, POD12-28). During endoscopies, the anastomosis will be lavaged with saline, the fluid will be collected by suction and images will be taken.
  Other Names: SES
Drug: Saline — During endoscopies after imaging, the anastomosis will be lavaged with a placebo direct topical saline solution
  Other Names: 0.9% saline solution
  Arms: Saline

SUMMARY:
Rationale: The surgical complication of intestinal anastomotic leak remains a clear and present danger to patients despite advances in surgical technique and ever more powerful antibiotics. No surgeon is immune from this complication and leak rates have not changed in decades. The consequences of a leak (peritonitis, sepsis, death) can be so severe that in the case of rectal cancer, diverting ileostomies are routinely performed to divert the fecal stream away from the healing anastomosis. We have recently discovered that certain intestinal bacteria, with the capacity to express collagenase and cleave MMP9 (Matrix metallopeptidase 9) to its active collagen degrading form, play a key and causative role in anastomotic leak. These bacteria often escape elimination due to the failure of current antibiotic regimens and their delivery methods to remain functionally durable at anastomotic tissue sites.

Purpose: This phase II clinical trial will track, in real time, the process of anastomotic healing and its associated microbiome by performing serial endoscopic surveillance (SES) following rectal cancer resection. By capturing anastomotic images and the associated microbial and inflammatory mediators from anastomotic fluids via SES performed at three time points following rectal cancer resection, we will correlate healing to microbial composition and inflammatory mediator status. Patients will be randomized and, at each time point, will receive lavage of their anastomosis with either saline or a triple antibiotic solution (ciprofloxacin, metronidazole, neomycin). An anastomotic healing score captured during SES will be compared between the two treatment arms and correlated to microbial and inflammatory mediator analyses of fluid samples to determine how intestinal microbes influence the process of anastomotic healing.

DETAILED DESCRIPTION:
OBJECTIVES

* Perform repeated postoperative endoscopy of anastomotic tissue sites in patients undergoing low anterior resection for rectal cancer with diverting ileostomy.
* Demonstrate that SES can reliably discriminate those anastomoses that progress along a continuum toward normal healing versus those that heal pathologically when images are evaluated by a jury blinded to treatment.
* Demonstrate that those anastomoses that are judged to progress pathologically harbor distinct microbial species and predictive inflammatory mediators.
* Demonstrate that when anastomotic tissues are lavaged with antibiotics directly via endoscopy (ciprofloxacin, metronidazole, neomycin), microbial pathogens that escape conventional antibiotics are eliminated and anastomotic healing progresses normally.
* Determine if the anastomotic healing score, microbial analyses, and/or inflammatory mediator analyses identify or predict symptomatic and clinically relevant anastomotic complications.

STUDY This is a randomized, multicenter study. All patients undergo resection of rectal cancer with a low anterior resection with anastomoses within 10cm of the anal verge and diverting ileostomy. Patients will undergo three endoscopies: one intra-operative endoscopy (POD0) and two post-operative endoscopies (POD3-7, POD12-28) (POD = post-operative day). During the SES procedure, the anastomosis will be lavaged with saline, the fluid will be collected by suction, images will be taken and then the anastomosis will be lavaged with either saline or an antibiotic solution composed of metronidazole, ciprofloxacin and neomycin. Patients' clinical courses will be followed through chart review for 6 to 7 months following surgery.

PROJECTED ACCRUAL A total of 200 patients (approximately 100 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of rectal cancer
* Scheduled to undergo a low anterior resection (with the planned anastomosis within 10cm of the anal verge) and a diverting ileostomy
* 18 years of age or older
* Able to provide informed consent

Exclusion Criteria

* Prior medical history of or suspected diagnosis of inflammatory bowel disease or irritable bowel syndrome
* Pregnant or breastfeeding
* Allergy to lidocaine, ciprofloxacin, metronidazole or neomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Anastomotic Healing Score (ordinal scale ranging from 0 to a maximum of 18) | Post-operative day 12-28

SECONDARY OUTCOMES:
Anastomotic Healing Score (ordinal scale ranging from 0 to a maximum of 18) | Post-operative day 0
Anastomotic Healing Score (ordinal scale ranging from 0 to a maximum of 18) | Post-operative day 3-7

CONTACTS AND LOCATIONS:
Overall Officials: John C Alverdy, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olivas AD, Shogan BD, Valuckaite V, Zaborin A, Belogortseva N, Musch M, Meyer F, Trimble WL, An G, Gilbert J, Zaborina O, Alverdy JC. Intestinal tissues induce an SNP mutation in Pseudomonas aeruginosa that enhances its virulence: possible role in anastomotic leak. PLoS One. 2012;7(8):e44326. doi: 10.1371/journal.pone.0044326. Epub 2012 Aug 31. PMID 22952955
- [Background] Shogan BD, Belogortseva N, Luong PM, Zaborin A, Lax S, Bethel C, Ward M, Muldoon JP, Singer M, An G, Umanskiy K, Konda V, Shakhsheer B, Luo J, Klabbers R, Hancock LE, Gilbert J, Zaborina O, Alverdy JC. Collagen degradation and MMP9 activation by Enterococcus faecalis contribute to intestinal anastomotic leak. Sci Transl Med. 2015 May 6;7(286):286ra68. doi: 10.1126/scitranslmed.3010658. PMID 25947163